CLINICAL TRIAL: NCT00306150
Title: A Multi-center, Randomized, Double Blind, Placebo Controlled Study to Investigate the Efficacy and Safety of Aprotinin on Transfusion Requirements in Patients With Bladder Cancer Undergoing Radical or Total Cystectomy.
Brief Title: Efficacy and Safety of Aprotinin on Transfusion Requirements in Patients Undergoing Radical or Total Cystectomy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12002; 2005-004055-35 (EudraCT Number)
Record Dates: First submitted 2006-03-21; First posted 2006-03-23 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Blood Loss, Surgical; Postoperative Hemorrhage
Keywords: Prevention of blood loss; Blood Loss, Surgical; Blood Loss, Postoperative
MeSH Terms: conditions — Blood Loss, Surgical; Postoperative Hemorrhage | interventions — Aprotinin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Trasylol (Aprotinin, BAYA0128)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trasylol (Aprotinin, BAYA0128) — Subjects will be randomized to receive an infusion of aprotinin (a test dose followed by a loading dose of 2 million KIU before skin incision followed by 500,000 KIU/hour until the end of surgery) or matching placebo. The maximal dose of aprotinin, that can be administered is 7,000,000 KIU, regardless of the duration of the operation. When a total of 7 million has been reached the administration of aprotinin must be discontinued.
  Arms: Arm 1
Drug: Placebo — Placebo is used according to the description of Arm 1
  Arms: Arm 2

SUMMARY:
The purpose of this study is to assess if aprotinin (BAYA0128), given intravenously during your surgery, is safe and can help reduce the need for a blood transfusion during bladder surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age and older
* Subjects requiring elective radical or total cystectomy for bladder cancer
* Documented, signed, dated informed consent obtained prior to any study specific procedures being performed

Exclusion Criteria:

* Subjects with previous exposure to aprotinin in the last 6 months or with a known or suspected allergy to aprotinin
* Subjects with sepsis or undergoing laparoscopic surgery
* Subjects with impaired renal function (serum creatinine >2.5 mg/dL or 221 micromoles/liter)
* Subjects with a history of bleeding diathesis, deep vein thrombosis or pulmonary embolism or known coagulation factor deficiency. Based on the investigator's opinion of any active significant medical illness the subject may have
* Subjects who refuse to receive allogenic blood products or whose preoperative red blood cell volume is so low that a blood transfusion would be likely to be given perioperatively (preoperative hematocrit of <24% or hemoglobin of <8 g/dl)
* Subjects who have participated in an investigational drug study within the past 30 days
* Subjects who are pregnant or breastfeeding or women of childbearing potential in whom the possibility of pregnancy cannot be excluded by a negative pregnancy test and who are not using a reliable method of contraception
* Planned use of other antifibrinolytic agents, e.g. aminocaproic acid or tranexamic acid
* Subjects on chronic anticoagulant treatment with warfarin that cannot be temporarily discontinued for the surgical procedure (as per local practices)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2005-12; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The primary criterion for efficacy is the percent of patients requiring a blood transfusion anytime in the intra-operative or post-operative period (up to the earlier of Day 7 or discharge) | Anytime in the intra-operative or post-operative period (up to the earlier of Day 7 or discharge)

SECONDARY OUTCOMES:
The number of units of blood or packed red cells transfused. There will be an analysis for the combination of autologous and allogenic transfusion and for allogenic alone | Intra- and postoperative
The number of units of blood or packed red cells transfused per patient requiring transfusion | Intra- and postoperative
The intraoperative blood loss determined as follow: a) by surgeon estimate b) summing weight of the blood in gauze and other materials and the suction drainage volume | Intraoperative
The drainage volume (in milliliters) from the operative site | In the first 8 hours post-operatively, and daily total drainage until removal of drains or until discharge, whichever comes first
Transfusion of platelets, colloids, plasma and number of patients requiring these products | Intra- and postoperative
The change from preoperative hemoglobin concentration to postoperative hemoglobin concentration | Obtained in the morning of postoperative Day 3, or, if transfused earlier, prior to transfusion
Surgeon s assessment of the degree to which bleeding obscures his/her view of the surgical field, relative to past, similar procedures | Intraoperative
Changes in blood markers related to inflammation and blood coagulation; baseline until Discharge or day 7 | Several measurements from baseline up to 6 weeks
Time to discontinuing of mechanical ventilation | Not specifed
Changes in FEV1 | Baseline until Discharge or day7
Changes in the patients health related quality of life (HRQoL) (at baseline and 6+-2 weeks post surgery) using the Functional Assessment Cancer Therapy for patients with Bladder cancer (FACT-Bl) questionnaire | At baseline and 6+-2 weeks post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (36):
- United States (17):
  - Los Angeles, California
  - Denver, Colorado
  - Miami, Florida
  - Chicago, Illinois
  - Portland, Maine
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - Rochester, Minnesota
  - Chapel Hill, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas
  - Burlington, Vermont
- Belgium (2):
  - Ghent
  - Leuven
- France (2):
  - Nantes
  - Nice
- Germany (7):
  - Tübingen, Baden-Wurttemberg
  - München, Bavaria
  - Regensburg, Bavaria
  - Fulda, Hesse
  - Mainz, Rhineland-Palatinate
  - Homburg, Saarland
  - Dresden, Saxony
- Netherlands (2):
  - Maastricht
  - Nijmegen
- Sweden (4):
  - Linköping
  - Lund
  - Stockholm
  - Uppsala
- United Kingdom (2):
  - Cambridge, Cambridgeshire
  - Newcastle upon Tyne, Tyne and Wear

REFERENCES:
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu